CLINICAL TRIAL: NCT03512236
Title: A Trial to Investigate Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of BioChaperone® Pramlintide Insulin in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CT031-ADO09
Record Dates: First submitted 2018-04-19; First posted 2018-04-30 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — pramlintide; Insulin, Regular, Human; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BC Pram Ins (Experimental): Single subcutaneous injection of BC Pram Ins + injection of placebo (0.9% NaCl) to ensure the double dummy
  Interventions: Drug: BC Pram Ins; Drug: Placebo
- Symlin® and Humulin® (Active Comparator): Simultaneous subcutaneous injections avec pramlintide and human insulin
  Interventions: Drug: Symlin® and Humulin®
- Humalog® (Active Comparator): Single subcutaneous injection of lispro + injection of placebo (0.9% NaCl) to ensure the double dummy
  Interventions: Drug: Humalog®; Drug: Placebo

INTERVENTIONS:
Drug: BC Pram Ins — Injection of BC Pram Ins
  Arms: BC Pram Ins
Drug: Symlin® and Humulin® — Injection of pramlintide and human insulin
  Arms: Symlin® and Humulin®
Drug: Humalog® — Injection of lispro
  Arms: Humalog®
Drug: Placebo — Injection of 0.9% NaCl
  Arms: BC Pram Ins; Humalog®

SUMMARY:
This is a single center, randomised, double-blind, active comparator controlled, three-period cross-over, single dose trial in subjects with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
This is a single center, randomised, double-blind, active comparator controlled, three-period cross-over, single dose trial in subjects with type 1 diabetes mellitus.

Each subject will be randomly allocated to a sequence of three treatments:(i) simultaneous administrations of BioChaperone® pramlintide human insulin (BC Pram Ins) and placebo, (ii) simultaneous injections of pramlintide (Symlin®) and human insulin (Humulin®) and (iii) simultaneous injections of insulin lispro (Humalog®) and placebo.

Subjects will come in a fasted state to the clinical trial centre in the morning, meal test procedures will be performed and subjects will stay at the clinical trial centre until the post-dose follow-up period has been terminated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-64 years (both inclusive)
* Type 1 diabetes mellitus (as diagnosed clinically) ≥ 12 months
* Treated with multiple daily insulin injections ≥ 12 months
* Treated with an evening dose of once-daily insulin glargine U100 at screening
* Fasting C-peptide ≤ 0.30 nmol/L

Exclusion Criteria:

* Known or suspected hypersensitivity to IMPs, paracetamol (acetaminophen) or related products
* Type 2 diabetes mellitus
* Clinically significant abnormal haematology, biochemistry, or urinalysis screening tests, as judged by the Investigator considering the underlying disease
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea), as judged by the Investigator
* Known slowing of gastric emptying, including gastroparesis, and or gastrointestinal surgery that in the opinion of the investigator might change gastrointestinal motility and food absorption
* Intake of medication known to affect gastrointestinal motility, including but not limited to erythromycin, metoclopramide, cisapride, cholestyramine or colestipol within 4 weeks before screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
CmaxPram | From 0 to 8 hours
  Maximum pramlintide concentration
AUCPram_0-8h | From 0 to 8 hours
  Area Under the pramlintide concentration-time Curve from 0-8 hours after IMP administration

SECONDARY OUTCOMES:
Pharmacokinetics of pramlintide | From 0 to 8 hours
  Area Under the pramlintide concentration-time Curve
Pharmacokinetics of insulins | From 0 to 8 hours
  Area Under the insulin concentration-time Curve
Glucose pharmacodynamics | From 0 to 8 hours
  Area Under the blood glucose concentration-time Curve
Safety and tolerability (Adverse Events recording) | From 0 to 8 hours
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: No